CLINICAL TRIAL: NCT07082439
Title: Phase II Trial of Pembrolizumab in Combination With Odetiglucan for Patients With Metastatic Colorectal Adenocarcinoma With Liver Predominant Disease
Brief Title: Pembrolizumab and Odetiglucan in Liver Predominant Metastatic Colorectal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05225
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Adenocarcinoma Metastatic in the Liver
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Odetiglucan (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Odetiglucan

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg intravenous administration on day 1 of each 3-week cycle until disease progression, unacceptable toxicity or participant withdrawal. Participants who complete study intervention after 2 years of pembrolizumab and odetiglucan without disease progression and subsequently experience disease progression while off of treatment are eligible for up to 1 year of additional pembrolizumab and odetiglucan (second course).
Drug: Odetiglucan — Odetiglucan 4 mg/kg intravenous administration on day 1 of each 3-week cycle until disease progression, unacceptable toxicity or participant withdrawal. Participants who complete study intervention after 2 years of pembrolizumab and odetiglucan without disease progression and subsequently experience disease progression while off of treatment are eligible for up to 1 year of additional pembrolizumab and odetiglucan (second course).

SUMMARY:
This study will evaluate the safety and effectiveness of the combination of pembrolizumab and odetiglucan in patients with metastatic colorectal cancer that is predominantly in the liver.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic colorectal adenocarcinoma with liver-predominant disease, defined as liver metastases with

  * No symptomatic lung or bony metastases
  * No peritoneal carcinomatosis or clinically significant ascites as determined by the investigator Note: at least 1 measurable lesion must be present in the liver to assess response. It is preferable to have at least 1 other lesion present in the liver which can be biopsied. Measurable lesions chosen as target lesions in the liver should not be biopsied if it can be avoided
* Patient must have received prior treatment with a fluoropyrimidine, oxaliplatin, irinotecan, and a VEGF inhibitor (e.g., bevacizumab), unless contraindicated.

  * Patients with KRAS/NRAS/BRAF wild-type cancers must also have received an EGFR inhibitor (e.g., cetuximab or panitumumab) in addition to the aforementioned therapies, unless contraindicated.
  * Patients who experienced disease recurrence within 6 months of oxaliplatin-containing adjuvant therapy will qualify as having received an oxaliplatin-containing regimen in the metastatic setting.
* Tumor must have documented mismatch repair proficiency (MMR proficient) by immunohistochemistry or not microsatellite instability high(non-MSI-H) by PCR.
* Participants who have adverse events due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy or persistent alopecia are eligible.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1 with at least one measurable lesion in the liver. It is preferable that one additional viable lesion in the liver that could be safely biopsied is also present, but not required for inclusion. Lesions chosen as target lesions in the liver should not be biopsied if possible. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Have a life expectancy of 3 months or greater as assessed by the investigator
* Have adequate organ function. Specimens must be collected within 14 days prior to the start of study intervention.
* Male participants: A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

* WOCBP who has a positive urine pregnancy test within 72 hours prior to receiving the first dose of study medication (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. If the serum pregnancy test is negative, then the participant will be deemed eligible on this criterion.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has previous treatment with odetiglucan
* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to first dose of study treatment.
* Has received prior radiotherapy within 2 weeks of start of study intervention or has ongoing radiation-related toxicities requiring corticosteroids.

  * Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease, with a 1-week washout, is permitted.
* Has undergone treatment chemoembolization or radioembolization within 6 weeks prior to enrollment on the study
* Has undergone hepatic arterial infusion pump placement
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Has received an investigational agent or has used an investigational device within the shorter of 4 weeks or 5 half-lives of the first dose of study intervention administration.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Note: No HIV testing is required unless mandated by local health authority.
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Hepatitis B and C screening tests are not required unless the participant has a known history of HBV and HCV infection. Participants may be eligible if the following criteria are met (18a and/or 18b).

  * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, have undetectable HBV viral load prior to initiation of study therapy, and should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention
  * Participants with history HCV infection are eligible if HCV viral load is undetectable at screening and have completed curative anti-viral therapy at least 4 weeks prior to randomization
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome within ≤ 6 months prior to start of study treatment, symptomatic or uncontrolled arrhythmia, congestive heart failure, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Proportion of patients with best response as complete response (CR) or PR (partial response) using RECIST v. 1.1.

SECONDARY OUTCOMES:
ORR iRECIST | Up to 2 years.
  Proportion of patients with best response of CR or PR as assessed by iRECIST.
ORR Liver by iRECIST | Up to 2 years.
  Proportion of patients with best response of CR or PR as assessed by iRECIST using only target lesions in the liver.
Duration of response | From date of first CR or PR by iRECIST until disease progression or death, whichever comes first, assessed up to 4 years.
  Time from first CR or PR by iRECIST to disease progression or death, whichever occurs first. Censoring will occur at the time of last patient contact if lost to follow-up, or at the time of data cutoff.
Disease control rate | Up to 2 years.
  Proportion of patients with PR, CR, or stable disease (SD) by iRECIST as best response.
Progression free survival | From date of enrollment to first documented disease progression or date of death from any cause, whichever came first, assessed up to 4 years.
  Time from enrollment to disease progression by iRECIST or death, whichever occurs first. Censoring will occur at the time of last patient contact if lost to follow-up, or at the time of data cutoff.
Overall survival | From date of enrollment to death from any cause assessed up to 4 years.
  Time from enrollment to death. Censoring will occur at the time of last patient contact if lost to follow-up, or at the time of data cutoff.
Toxicity rates | Will be assessed during the adverse event reporting period from the initiation of study intervention through 30 days following cessation of study intervention.
  Toxicity rates will be assessed as an ordinal measure (e.g., Grade 1 pneumonitis, Grade 2 pneumonitis, etc.) using CTCAE v. 5.0. Toxicity rates will be summarized as a proportion of patients experiencing each toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: William Chapin, MD, MSCE, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the clinical trial publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months following clinical trial publication. No end date.
Access Criteria: To achieve aims in an approved proposal. Proposals should be directed to corresponding author on the clinical trial publication.